## Title: Group ("Project Life Force") vs. Individual Suicide Safety Planning RCT

NCT Number: NCT03653637

Date: 05/12/2025

## Primary Statistical Analysis Plan

The primary outcome of suicidal behavior will be analyzed using a Cox Proportional Hazard Regression, with treatment condition (PLF+TAU vs. TAU) and baseline suicidal behavior level as predictors, and incidence and time to the first suicidal behavior during the study course as the outcome variables. The model will adjust for treatment site. Kaplan-Meier estimates of the cumulative hazard function for both groups will be graphed and the proportionality assumption checked. If the hazard functions are not proportional, the non-parametric log-rank test will be used instead, with treatment condition as predictor, and we will use a sensitivity analysis to test the effect of baseline suicidal behavior severity by splitting the treatment conditions by the presence/absence suicidal behavior.

Most secondary and other outcomes (depression, hopelessness, thwarted belongingness, aggression dimensions, insomnia and suicide-related coping) will be analyzed in Linear Mixed Effects (LME) regression models. All LMEs will be adjusted for site and will include randomization condition, time, and a randomization by time interaction. The treatment effect of PLF+TAU vs TAU will be the treatment by time interaction. Time will be treated as a linear variable. Mixed-effect models can be fit to data with dropout or missing values as long as the data is missing at random, thus, attrition does not necessarily reduce the number of participants included in these analyses.

For the two outcomes (drug and alcohol use) that are only measured at the one-year follow-up (with retrospective questions about the past 12 months), we will compare between PLF+TAU and TAU with t-tests or Mann-Whitney U tests where appropriate.